CLINICAL TRIAL: NCT04693806
Title: The Effect of Embryo Culture Under a Continuous CO2 Setting Versus a Sequential CO2 Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RMA-2020-04
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous CO2 Level (Experimental): embryos will remain in a single incubator set at a continuousCO2 level
  Interventions: Other: Continuous CO2 Level
- Sequential CO2 Level (No Intervention): Current standard of care

INTERVENTIONS:
Other: Continuous CO2 Level — Embryos will be cultured in a single, continuous CO2 setting
  Arms: Continuous CO2 Level

SUMMARY:
The purpose of this study is to determine if embryo culture under a single CO2 setting improves blastocyst formation rate.

DETAILED DESCRIPTION:
Following enrollment, patients will undergo ovarian stimulation and oocyte retrieval per routine as previously consented to at the clinic. IVF stimulation protocol will be at the discretion of the patient's individual provider, per routine. Intracytoplasmic Sperm Injection (ICSI) will be performed and embryos will be cultured to the blastocyst stage per routine. There are no changes to the embryology care itself, the only difference within the study is the CO2 level within the incubator pending the patient's randomization.

ELIGIBILITY:
Major Inclusion Criteria for participants:

1. Patients undergoing IVF stimulation cycle with plan for subsequent FET

Major Exclusion Criteria for participants:

1. All patients who do not voluntarily give their written consent for participation
2. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
3. Use of surgical procedures to obtain sperm

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
blastulation rate | approximately one week
  the number of zygotes that reach the blastocyst stage

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No